CLINICAL TRIAL: NCT01153451
Title: An Automatic Notification System for Test Results Finalized After Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anuj K. Dalal, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R21HS018229-01 (AHRQ); CRICO (Other Grant/Funding Number: CRICO)
Record Dates: First submitted 2010-06-03; First posted 2010-06-30 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Test Result Management
Keywords: Pending tests; Discharge; Awareness; Care transitions

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Responsible inpatient and ambulatory physicians assigned to usual care will not receive any email(s) of patients' test results generated from the notification system.
- Email Notification (Other): Responsible inpatient and ambulatory physicians will receive automated email(s) of patients' tests results finalized post-discharge generated from the notification system. Finalized results will be batched such that no provider will receive more than one email per day.
  Interventions: Other: Email Notification

INTERVENTIONS:
Other: Email Notification — BWH inpatient clinical information systems will automatically file all non-finalized chemistry, hematology, pathology, and radiology tests, as well as inpatient and ambulatory provider email addresses for all study patients discharged. This process will be initiated using a time stamp most proximate to actual discharge time. At midnight on every day, all tests filed at time of discharge will be updated if final results have become available. An email with all finalized and pending test results for each patient discharged will be sent to the inpatient and primary care provider at this time. For patients discharged with more than one pending test, subsequent email notification(s) will be sent out until all pending tests are finalized (no more than one email per day).
  Arms: Email Notification

SUMMARY:
Specific Aims: (Study #1, funded by AHRQ, completed May 2011)

1. To create an automatic notification system to prompt physicians of test results finalized after discharge.
2. To evaluate the impact of this system on physician awareness of test results finalized after discharge.

Hypothesis: Automatic email notification will improve physician awareness of test results finalized after discharge compared to usual care.

Specific Aims: (Study #2, funded by CRICO, completed July 2012)

1. To identify a cohort of discharged patients with potentially actionable results of tests pending at discharge (TPAD).
2. To determine if automated email notification of the finalized results of potentially actionable TPADs affects the rate of post-discharge actions taken as documented in the electronic medical record (EMR).

Hypothesis: Automated email notification of the finalized results of potentially actionable TPADs increases the rate of actions taken post-discharge.

DETAILED DESCRIPTION:
Failure to follow up on abnormal test results is a critical problem and is more likely to occur in the case of tests that are performed in the hospital but whose results are not available or not finalized until after discharge (i.e., pending test results). Responsible inpatient and ambulatory providers may not be aware of these test results. In a prior study, Roy et al. determined that 41% of patients were discharged before all laboratory, microbiology, and radiology test results were finalized (31% were collectively hematology, chemistry, and pathology tests, 27% were radiology studies, and 42% were microbiology results). Of these results, 9.4% were considered potentially actionable by independent physician review and could have altered the post-discharge patient care plan. Physicians were only aware of 38% of these test results. Failure to follow-up on these test results can lead to delays in diagnosis, missed treatment opportunities, redundant ordering of tests, and subsequent patient harm. In a hospital the size of Brigham and Women's Hospital (BWH) with 44,000 annual admissions, physicians would be unaware of almost 2000 actionable test results per year. Automated systems can mitigate this problem by ensuring prompt notification of relevant test results finalized after discharge to responsible inpatient and ambulatory providers. Using internal BWH funding, we have developed an automated email notification system to facilitate management of tests pending at discharge (TPADs).

In study 1 (funded by AHRQ), we will prospectively evaluate the impact of this intervention on physician awareness of TPAD results. In study 2 (funded by CRICO), we will perform a chart review to determine the impact of the intervention on downstream actions taken by physicians and acknowledgment of TPAD results as documented in the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Any patient discharged from selected services at BWH whose inpatient attending and primary care provider are in the same arm of the study.

Exclusion Criteria:

* Any patient discharged from selected services at BWH whose inpatient attending and primary care provider are in discordant arms of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percent of Inpatient Providers Aware of Finalized Results of Tests Pending at Discharge (Study 1) | 72 hours after notification, October 2010 thru May 2011
  The primary outcome will be the percentage of inpatient physicians who are aware of the finalized results of tests pending at discharge.

SECONDARY OUTCOMES:
Percent of Ambulatory Providers Aware of Finalized Results of Tests Pending at Discharge (Study 1) | 72 hours after notification, October 2010 thru May 2011
  Secondary outcomes will include the percentage of ambulatory physicians who are aware of the finalized results of tests pending at discharge (both Partners network and non-network providers).
Percent of Providers Aware of Actionable Test Results (Study 1) | 72 hours after notification, October 2010 thru May 2011
  Percent awareness of actionable test results by responsible providers
Provider Satisfaction (Study 1) | 72 hours after notification, October 2010 thru May 2011
  Percentage of providers satisfied with the notification system.

OTHER OUTCOMES:
Proportion of potentially actionable TPAD results with documented action(s) taken in the intervention versus control arms. (Primary Outcome, Study 2) | Retrospective chart data abstraction for patients discharged from July 2011 through July 2012
  The primary outcome will be measured as the difference in the proportion of potentially actionable TPAD results with documented actions taken (as determined by electronic chart review) per discharged patient in the intervention and control arm.
Proportion of potentially actionable TPAD results with documented acknowledgement in the intervention versus control arms. (Secondary Outcome, Study 2) | Retrospective chart data abstraction for patients discharged from July 2011 through July 2012
  The secondary outcome will be measured as the difference in the proportion of potentially actionable TPAD results with documented acknowledgment (as determined by electronic chart review) in the intervention and control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anuj K Dalal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Dalal AK, Schaffer A, Gershanik EF, Papanna R, Eibensteiner K, Nolido NV, Yoon CS, Williams D, Lipsitz SR, Roy CL, Schnipper JL. The Impact of Automated Notification on Follow-up of Actionable Tests Pending at Discharge: a Cluster-Randomized Controlled Trial. J Gen Intern Med. 2018 Jul;33(7):1043-1051. doi: 10.1007/s11606-018-4393-y. Epub 2018 Mar 12. PMID 29532297
- [Derived] Dalal AK, Roy CL, Poon EG, Williams DH, Nolido N, Yoon C, Budris J, Gandhi T, Bates DW, Schnipper JL. Impact of an automated email notification system for results of tests pending at discharge: a cluster-randomized controlled trial. J Am Med Inform Assoc. 2014 May-Jun;21(3):473-80. doi: 10.1136/amiajnl-2013-002030. Epub 2013 Oct 23. PMID 24154834